CLINICAL TRIAL: NCT05216536
Title: Better Understanding Physical and Cognitive Impairments and Functional Limitations in People Suffering From Long COVID to Support the Development of Adapted Interventions
Brief Title: Physical and Cognitive Impairments in People Suffering From Long COVID
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-2328
Record Dates: First submitted 2022-01-14; First posted 2022-01-31 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; SARS-CoV-2 Infection; Corona Virus Infection; Physical Disability; Cognitive Impairment; Cognitive Dysfunction; Quality of Life; Symptoms and Signs; Impairment
Keywords: Long covid; Long-haul; Chronic; Post-acute; Sequelae; Persistent; Physical health; Physical fitness; Function; Limitation; Health-related quality of life
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Cognitive Dysfunction; Signs and Symptoms; Post-Acute COVID-19 Syndrome; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Long COVID: Adults who contracted COVID-19 and present at least one physical or cognitive long COVID-19 symptom for more than 12 weeks following the initial diagnosis.
  Interventions: Other: No intervention
- Acute COVID: Adults who contracted COVID-19 but did not experience persistent symptoms for more than 4 weeks following the initial diagnosis.
  Interventions: Other: No intervention
- Control: Adults who did not contract COVID-19.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Of the 1,900,000 Canadians who have been infected by COVID-19, 8 to 15% will continue to experience COVID-19 related symptoms well after 12 weeks. The persistence of such symptoms is now defined as "long COVID" syndrome. Current evidence does not provide a clear understanding of the physical and cognitive impairments and functional limitations that persons with long COVID present. The objectives of this project are to describe the physical and cognitive impairments and functional limitations experienced by people with long COVID and compare the evolution over 6 months of people from three separate groups: a group of people with long COVID (long COVID Group), another group of people who contracted COVID-19 but did not experience persistent symptoms (acute COVID Group), and a group of people who did not contract COVID-19 (Control Group).

One hundred and twenty adults in each of the three groups will be recruited and will take part in three evaluations within 6 months (baseline and 3 and 6 months after baseline). At baseline, all participants will complete questionnaires on sociodemographics, COVID symptomatology and comorbidity, and self-reported questionnaires on quality of life, functional status, sleep, pain-related disabilities, anxiety, depression, fatigue and cognitive function. Then, physical and cognitive tests will be performed in a laboratory to provide complementary results on impairments and functional limitations. Finally, participants will wear a fitness tracker watch to monitor their activity and sleep for 7 days. The participants will complete the same measures (questionnaires, lab measures, fitness tracker watch) at 3 and 6 months after baseline evaluations.

This project will lead to a better understanding of the impairments/limitations experienced following COVID-19. Hence, these results will allow to identify the interventions needed by the population and ensure these are offered through effective healthcare pathways.

DETAILED DESCRIPTION:
The objectives of this study are to: describe the physical and cognitive impairments and functional limitations experienced by individuals with long COVID using self-reported and objective clinical measures and compare the evolution over time of the physical and cognitive state and level of functioning between: a) people with long COVID, b) people who contracted COVID-19 but did not experience persistent symptoms, and c) people who did not contract COVID-19.

One hundred and twenty adults with long COVID symptoms (Long COVID Group), 120 age- and sex-matched adults who contracted COVID-19 but did not experience persistent symptoms (Acute COVID Group) and 120 age- and sex-matched adults who did not contract COVID-19 (Control Group) will take part in three evaluations within 6 months (baseline and 3 and 6 months after baseline). The baseline evaluation will include 1) the completion of web-based self-administered questionnaires (quality of life, functional status, sleep, pain-related disabilities, anxiety, depression, fatigue and cognitive function); 2) an in-lab session at one of the two participating research centers (Centre interdisciplinaire de recherche en réadaptation et en intégration sociale [Cirris] in Quebec City, Centre de recherche de l'Hôpital Maisonneuve-Rosemont [CRHMR] in Montreal) during which participants will answer questions on sociodemographics, COVID-19 medical history and symptoms experienced, and will perform clinical tests to objectify cognitive and physical impairments and functional limitations (attention, memory, executive functioning, grip strength, balance, gait speed and endurance, oxygen consumption [VO2] and metabolic cost of walking), and 3) wearing a fitness tracker watch to monitor activity and sleep for 7 days. The participants will complete the same measures (questionnaires, lab measures, fitness tracker watch) at three and 6 months after baseline evaluation

Statistical analyses for objective 1 will aim at presenting a sociodemographic and COVID history profiles of the Long COVID Group at baseline according to sex, gender, hospitalization, time since onset and comorbidities. Scores at baseline on self-reported and clinical variables will also be compared with the Acute COVID and Control Groups via three-group One-way ANOVA (maximum-likelihood ANOVA). For objective 2, repeated measures ANOVA will be used to compare the divergence in longitudinal performance across groups in self-reported and clinical variables (generalized ANOVA for repeated measures).

Gaining a greater understanding of the physical and cognitive state and level of functioning of persons with long COVID and on characteristics of those who will have a poorer outcome will help better define healthcare needs of these persons and guide the development of appropriate medical and rehabilitation interventions. Best practices in terms of medical and rehabilitation services in cases of long COVID are still just emerging and offering appropriate services to persons suffering from long COVID may contribute to improving outcomes such as long-term physical and cognitive impairments and functional limitations, as well as health-related quality of life.

ELIGIBILITY:
Inclusion Criteria

* For all 3 groups: 18 years of age or older and being able to participate in 3 evaluation sessions within 6 months
* For the COVID Groups: having received a diagnosis of COVID-19 from a government designated testing clinic or hospital at least 12 weeks prior to inclusion.
* For the Long COVID Group: presenting at least one physical or cognitive long COVID-19 symptom for more than 12 weeks following the initial diagnosis such as fatigue, shortness of breath, muscle weakness, joint pain, headache, cognitive dysfunction, or sleep-related difficulties
* For the Acute COVID Group: not have experienced any persistent symptom for more than 4 weeks after having contracted COVID- 19
* For the Control Group: not have received a diagnosis of COVID-19 and not have experienced COVID-19 symptoms since February 2020 such as fever, sudden loss of smell, headache, dyspnea, great fatigue, muscle or body aches, shortness of breath or sore throat

Exclusion criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred and twenty adults with long COVID symptoms (long COVID Group), 120 age- and sex-matched adults who contracted COVID-19 but did not experience persistent symptoms (acute COVID Group) and 120 age- and sex-matched adults who did not contract COVID-19 (Control Group) will be recruited through medical clinics in Quebec City and Montreal (e.g., Academic family medicine groups [FMG-U] and long COVID Clinics), invitations in newsletters sent to healthcare workers of CIUSSS de la Capitale-Nationale and CIUSSS de l'Est-de-l'Île-de-Montréal, electronic mailing lists of students, employees and retired employees at Université Laval (> 52,000 individuals), and social media (Facebook®, Instagram®).
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) baseline | Baseline
  5-level EQ-5D (EQ-5D-5L): generic HRQoL self-reported questionnaire that contains 5 questions covering 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Health-related quality of life (HRQoL) at 3 months | 3-month follow-up
  5-level EQ-5D (EQ-5D-5L): generic HRQoL self-reported questionnaire that contains 5 questions covering 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Health-related quality of life (HRQoL) at 6 months | 6-month follow-up
  5-level EQ-5D (EQ-5D-5L): generic HRQoL self-reported questionnaire that contains 5 questions covering 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression

SECONDARY OUTCOMES:
Comorbidities | Baseline
  Self- Administered Comorbidity Questionnaire (SCQ): generic questionnaire with 13 common medical conditions.
Sleep Quality | Baseline
  Pittsburgh Sleep Quality Index (PSQI): evaluates the quality and patterns of sleep over the last month.
Sleep Quality | 3-month follow-up
  Pittsburgh Sleep Quality Index (PSQI): evaluates the quality and patterns of sleep over the last month.
Sleep Quality | 6-month follow-up
  Pittsburgh Sleep Quality Index (PSQI): evaluates the quality and patterns of sleep over the last month.
Pain & Pain-Related Disabilities | Baseline
  Brief Pain Inventory Short Form (BPI-SF): designed to evaluate the intensity of, and the impairment caused by pain.
Pain & Pain-Related Disabilities | 3-month follow-up
  Brief Pain Inventory Short Form (BPI-SF): designed to evaluate the intensity of, and the impairment caused by pain.
Pain & Pain-Related Disabilities | 6-month follow-up
  Brief Pain Inventory Short Form (BPI-SF): designed to evaluate the intensity of, and the impairment caused by pain.
Anxiety | Baseline
  General Anxiety Disorder (GAD-7): assesses the seven core symptoms of generalized anxiety disorder by asking how frequent participants have been bothered by symptoms of anxiety.
Anxiety | 3-month follow-up
  General Anxiety Disorder (GAD-7): assesses the seven core symptoms of generalized anxiety disorder by asking how frequent participants have been bothered by symptoms of anxiety.
Anxiety | 6-month follow-up
  General Anxiety Disorder (GAD-7): assesses the seven core symptoms of generalized anxiety disorder by asking how frequent participants have been bothered by symptoms of anxiety.
Depressive symptoms | Baseline
  Patient-Health Questionnaire (PHQ-9): assesses the nine symptoms of a major depressive episode.
Depressive symptoms | 3-month follow-up
  Patient-Health Questionnaire (PHQ-9): assesses the nine symptoms of a major depressive episode.
Depressive symptoms | 6-month follow-up
  Patient-Health Questionnaire (PHQ-9): assesses the nine symptoms of a major depressive episode.
Fatigue | Baseline
  Fatigue Severity Scale (FSS): measures the severity of fatigue and its effect on a person's activities and lifestyle
Fatigue | 3-month follow-up
  Fatigue Severity Scale (FSS): measures the severity of fatigue and its effect on a person's activities and lifestyle
Fatigue | 6-month follow-up
  Fatigue Severity Scale (FSS): measures the severity of fatigue and its effect on a person's activities and lifestyle
Self-reported cognitive function | Baseline
  Patient Reported Outcomes Measurement Information System (PROMIS): the PROMIS Short Form v2.0 - Cognitive Function measures perceived changes in cognitive function.
Self-reported cognitive function | 3-month follow-up
  Patient Reported Outcomes Measurement Information System (PROMIS): the PROMIS Short Form v2.0 - Cognitive Function measures perceived changes in cognitive function.
Self-reported cognitive function | 6-month follow-up
  Patient Reported Outcomes Measurement Information System (PROMIS): the PROMIS Short Form v2.0 - Cognitive Function measures perceived changes in cognitive function.
Persistent symptoms | Baseline (long COVID group only)
  Newcastle post-COVID syndrome Follow Up Screening Questionnaire: identifies individuals who are experiencing residuals COVID-19 related symptoms and for who multi-disciplinary management or specialist support may be beneficial.
Persistent symptoms | 3-month follow-up (long COVID group only)
  Newcastle post-COVID syndrome Follow Up Screening Questionnaire: identifies individuals who are experiencing residuals COVID-19 related symptoms and for who multi-disciplinary management or specialist support may be beneficial.
Persistent symptoms | 6-month follow-up (long COVID group only)
  Newcastle post-COVID syndrome Follow Up Screening Questionnaire: identifies individuals who are experiencing residuals COVID-19 related symptoms and for who multi-disciplinary management or specialist support may be beneficial.
Cognitive function - MoCA | Baseline
  MoCA: assesses short term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language and orientation in time and place.
Cognitive function - MoCA | 3-month follow-up
  MoCA: assesses short term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language and orientation in time and place.
Cognitive function - MoCA | 6-month follow-up
  MoCA: assesses short term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language and orientation in time and place.
Cognitive function - auditory attention and working memory | Baseline
  Digit Span subtest of the WAIS-IV battery (including forward and Backward tasks): assesses auditory attention and working memory.
Cognitive function - auditory attention and working memory | 3-month follow-up
  Digit Span subtest of the WAIS-IV battery (including forward and Backward tasks): assesses auditory attention and working memory.
Cognitive function - auditory attention and working memory | 6-month follow-up
  Digit Span subtest of the WAIS-IV battery (including forward and Backward tasks): assesses auditory attention and working memory.
Cognitive function - information processing and executive functioning | Baseline
  Trail Making Test: assesses speed of information processing and executive functioning.
Cognitive function - information processing and executive functioning | 3-month follow-up
  Trail Making Test: assesses speed of information processing and executive functioning.
Cognitive function - information processing and executive functioning | 6-month follow-up
  Trail Making Test: assesses speed of information processing and executive functioning.
Grip strength | Baseline
  Grip Strength: Grip strength of both hands will be measured using a handgrip dynamometer. Grip strength is associated with concurrent overall strength, upper limb function and quality of life. Three trials will be performed, and the maximum strength reached will be used in the subsequent analysis.
Grip strength | 3-month follow-up
  Grip Strength: Grip strength of both hands will be measured using a handgrip dynamometer. Grip strength is associated with concurrent overall strength, upper limb function and quality of life. Three trials will be performed, and the maximum strength reached will be used in the subsequent analysis.
Grip strength | 6-month follow-up
  Grip Strength: Grip strength of both hands will be measured using a handgrip dynamometer. Grip strength is associated with concurrent overall strength, upper limb function and quality of life. Three trials will be performed, and the maximum strength reached will be used in the subsequent analysis.
Lower extremity function (including balance, gait speed and lower extremity strength) | Baseline
  Short performance physical battery (SPPB): The SPPB is a short (5-10 min) test to measure lower extremity function using tasks that mimic daily activities. It examines 3 areas of lower extremity function, including static standing balance (3 timed standing positions), gait speed (time to complete 4m walk), and getting in and out of a chair (time to complete 5x sit to stand).
Lower extremity function (including balance, gait speed and lower extremity strength) | 3-month follow-up
  Short performance physical battery (SPPB): The SPPB is a short (5-10 min) test to measure lower extremity function using tasks that mimic daily activities. It examines 3 areas of lower extremity function, including static standing balance (3 timed standing positions), gait speed (time to complete 4m walk), and getting in and out of a chair (time to complete 5x sit to stand).
Lower extremity function (including balance, gait speed and lower extremity strength) | 6-month follow-up
  Short performance physical battery (SPPB): The SPPB is a short (5-10 min) test to measure lower extremity function using tasks that mimic daily activities. It examines 3 areas of lower extremity function, including static standing balance (3 timed standing positions), gait speed (time to complete 4m walk), and getting in and out of a chair (time to complete 5x sit to stand).
Gait endurance | Baseline
  6-minute walk test (6MWT): The 6MWT will be performed in a 15 to 20-meter corridor and the distance covered will be measured with a measuring wheel.
Gait endurance | 3-month follow-up
  6-minute walk test (6MWT): The 6MWT will be performed in a 15 to 20-meter corridor and the distance covered will be measured with a measuring wheel.
Gait endurance | 6-month follow-up
  6-minute walk test (6MWT): The 6MWT will be performed in a 15 to 20-meter corridor and the distance covered will be measured with a measuring wheel.
Oxygen consumption (VO2) | Baseline
  Oxygen consumption (VO2) will be measured during the 6WMT using indirect calorimetry collected by a portable gas analysis system (Metamax® 3b).
Oxygen consumption (VO2) | 3-month follow-up
  Oxygen consumption (VO2) will be measured during the 6WMT using indirect calorimetry collected by a portable gas analysis system (Metamax® 3b).
Oxygen consumption (VO2) | 6-month follow-up
  Oxygen consumption (VO2) will be measured during the 6WMT using indirect calorimetry collected by a portable gas analysis system (Metamax® 3b).
Metabolic cost of walking | Baseline
  Metabolic cost of walking will be measured during the 6WMT using indirect calorimetry collected by a portable gas analysis system (Metamax® 3b).
Metabolic cost of walking | 3-month follow-up
  Metabolic cost of walking will be measured during the 6WMT using indirect calorimetry collected by a portable gas analysis system (Metamax® 3b).
Metabolic cost of walking | 6-month follow-up
  Metabolic cost of walking will be measured during the 6WMT using indirect calorimetry collected by a portable gas analysis system (Metamax® 3b).
Frailty | Baseline
  Clinical Frailty Scale (CFS): The CFS is a scale used to grade frailty and thus, identify participants who are at a higher risk of poor outcomes.
Frailty | 3-month follow-up
  Clinical Frailty Scale (CFS): The CFS is a scale used to grade frailty and thus, identify participants who are at a higher risk of poor outcomes.
Frailty | 6-month follow-up
  Clinical Frailty Scale (CFS): The CFS is a scale used to grade frailty and thus, identify participants who are at a higher risk of poor outcomes.
Physical activity - Number of steps in real-life environment | Baseline
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The average daily number of steps will be retrieved
Physical activity - Number of steps in real-life environment | 3-month follow-up
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The average daily number of steps will be retrieved
Physical activity - Number of steps in real-life environment | 6-month follow-up
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The average daily number of steps will be retrieved
Physical activity - Weekly number of minutes of moderate and intense activity in real-life environment | Baseline
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations.The weekly number of minutes of moderate and intense activity will be retrieved
Physical activity - Weekly number of minutes of moderate and intense activity inreal-life environment | 3-month follow-up
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations.The weekly number of minutes of moderate and intense activity will be retrieved
Physical activity - Weekly number of minutes of moderate and intense activity in real-life environment | 6-month follow-up
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations.The weekly number of minutes of moderate and intense activity will be retrieved
Sleep: Sleep time in real-life environment | Baseline
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The sleep time will be retrieved from the fitness tracker watch
Sleep: Sleep time in real-life environment | 3-month follow-up
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The sleep time will be retrieved from the fitness tracker watch
Sleep: Sleep time in real-life environment | 6-month follow-up
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The sleep time will be retrieved from the fitness tracker watch
Sleep: Sleep efficiency in real-life environment | Baseline
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The sleep efficiency will be retrieved from the fitness tracker watch
Sleep: Sleep efficiency in real-life environment | 3-month follow-up
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The sleep efficiency will be retrieved from the fitness tracker watch
Sleep: Sleep efficiency in real-life environment | 6-month follow-up
  Participants will be asked to wear a fitness tracker watch (Garmin Forerunner 35) 24 hrs/day for 7 consecutive days after each of the three physical evaluations. The sleep efficiency will be retrieved from the fitness tracker watch

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PT, PhD, Principal Investigator — Laval University
Locations (1):
- Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zahouani I, Desmeules F, Perreault K, Campeau-Lecours A, Best K, Beaulieu-Bonneau S, Paquette JS, Deslauriers S, Daigle N, Drouin G, Tittley J, Gagnon MA, Salmam I, Brouillard SM, Lepage K, Roy JS. Physical and cognitive impairments in people suffering from long COVID: protocol for a longitudinal population-based cohort study. BMJ Open. 2023 Mar 15;13(3):e064054. doi: 10.1136/bmjopen-2022-064054. PMID 36921943